CLINICAL TRIAL: NCT06961448
Title: A Prospective, Multi-center, Evaluator-blinded, Randomized, Parallel-controlled, Superiority Clinical Trial to Evaluate the Safety and Efficacy of Polycaprolactone Microsphere Fillers for Correction of Moderate to Severe Nasolabial Folds
Brief Title: A Study in Adults Evaluating Polycaprolactone Microsphere Filler for Treatment of Moderate to Severe Nasolabial Folds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Collaborators: Hangzhou Inshow Biotechnology Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LF30_NLF_China
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Nasolabial Fold Correction
Keywords: Polycaprolactone microsphere filler; Nasolabial folds
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyaluronate Gel for Injection (Active Comparator): HA filler
  Interventions: Device: Hyaluronate Gel for Injection
- Lafullen (Experimental): PCL filler
  Interventions: Device: Polycaprolactone microsphere filler

INTERVENTIONS:
Device: Hyaluronate Gel for Injection — Apply a maximum of 1.5 mL per side of the nasolabial fold using the test device (Lafullen) or the control device, with an optional touch-up of up to 0.5 mL per side at 4 weeks based on investigator assessment.
  Arms: Hyaluronate Gel for Injection
Device: Polycaprolactone microsphere filler — Apply a maximum of 1.0 mL per side of the nasolabial fold using the test device (Lafullen) or the control device, with an optional touch-up of up to 0.5 mL per side at 4 weeks based on investigator assessment.
  Arms: Lafullen

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of polycaprolactone microsphere filler (Lafullen) for the correction of moderate to severe nasolabial folds in adults aged 18 and above, regardless of gender.

The main questions it aims to answer are:

* Does Lafullen improve wrinkle severity in the nasolabial fold area at 48 weeks post-injection (WSRS responder rate)?
* Is Lafullen superior to the control product (Restylane, a hyaluronic acid filler) in terms of long-term wrinkle correction and safety? Researchers will compare Lafullen (polycaprolactone filler) with Restylane (modified sodium hyaluronate gel) to see if Lafullen provides superior wrinkle correction at 12 months post-injection.

Participants will:

* Receive either Lafullen or Restylane via injection in the nasolabial fold area.
* Optionally receive a touch-up injection at 4 weeks after the first treatment if needed.
* Undergo regular follow-up visits at 4, 12, 24, 36, and 48 weeks post-treatment.
* Subjects in the Lafullen group will continue follow-up up to 72 weeks to assess long-term efficacy and safety.
* Be assessed through clinical photography, pain scale (VAS), satisfaction questionnaires, and safety evaluations (e.g., AEs, vital signs, lab tests).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above, with no gender restriction.
2. Willing to receive treatment for correcting nasolabial fold.
3. Treatment investigator evaluate those with a WSRS score of 3 or 4 for bilateral nasolabial folds;
4. Willing to voluntarily participate in the clinical trial, accepting the obligation not toreceive all plastic surgery and cosmetic dermatology procedures or treatments during the trial。 Willing and able to undergo the required treatment and follow-up observations, and sign the informed consent form.

Exclusion Criteria:

1. Allergy to polycaprolactone, hyaluronic acid products or any component of the investigational device or control device(such as streptococcal proteins), allergy to any local anesthetic (such as lidocaine or other amide-typeanesthetic), or history of severe allergic reactions and multiple severe allergic reactions.
2. Previous surgery, cosmetic facial procedure, or plans to undergo cosmetic surgery in NLF area or lower face during the trial, inculding any of the following circumstances:

   1. Received permanent fillers or prostheses (such as PMMA etc.) or semi-permanent dermal fillers (such as CaHA, PLLA, PCL, etc.).
   2. Received temporary dermal fillers (such as HA and collagen etc.) within 12 months prior to screening.
   3. Received anti-wrinkle surgery within 12 months prior to screening.
   4. Receiving botulinum toxin injection, chemical stripping, radiofrequency laser, and liquid nitrogen freezing anti-wrinkle treatment within 6 months.
3. Individuals who used topical agents (e.g., corticosteroids, steroids [excluding hydrocortisone], retinoids, or retinoid derivatives intended as medications but not as cosmetics) on the mid-to-lower facial area within 3 months prior to screening or plan to use them during the trial period, as well as those undergoing hydrocortisone treatment.
4. Individuals with abnormal coagulation mechanisms [activated partial thromboplastin time (APTT) >1.5 times the upper limit of normal (ULN), etc.], or use of anticoagulants (e.g., warfarin, rivaroxaban), antiplatelet agents (e.g., aspirin, clopidogrel), thrombolytic agents (e.g., recombinant human urokinase) within 2 weeks prior to screening.
5. Individuals with severe liver or kidney dysfunction, such as liver function markers (ALT, AST) exceeding 2 times the ULN or kidney function markers (creatinine) exceeding 1.5 times the ULN.
6. Individuals with infectious diseases, including any positive test results for hepatitis B surface antigen, hepatitis C antibodies, HIV antibodies, or syphilis antibodies.
7. Individuals with scars, unhealed wounds, deformities, defects, tattoos, or excessive pigmentation in the nasolabial fold area that may affect the efficacy assessment.
8. Individuals with tumors, precancerous lesions, active skin lesions such as herpes, in the nasolabial fold area.
9. Individuals with acute or chronic skin diseases such as infections or inflammation in the treatment area.
10. Individuals with autoimmune diseases, such as psoriasis.
11. Individuals with uncontrolled diabetets.
12. Individuals prone to scarring, keloid formation, or hypertrophic scars.
13. Individuals diagnosed with psychiatric disorders, lacking self-autonomy, or experiencing active episodes of anxiety or depression.
14. Individuals with excessively high expectations of treatment outcomes or unwilling to accept potential short-term side effects such as bruising, swelling, or pain.
15. Individuals who are pregnant, breastfeeding, or unwilling to use medically approved contraception (e.g., oral contraceptives, condoms, intrauterine devices) during the trial.
16. Individuals who participated in other drug or medical device clinical trials within 3 months prior to screening.
17. Individuals deemed unsuitable for trial participation by the investigator for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
WSRS Responder Rate at Week 48 | 48 weeks after injection
  Wrinkle Severity Rating Scale (WSRS) responder rate: Percentage of participants showing ≥1-point improvement from baseline in WSRS on both sides of the nasolabial folds, as evaluated by a blinded assessor using standardized facial photographs. A higher percentage indicates greater wrinkle correction efficacy.

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) has not been finalized. While we recognize the potential value of IPD sharing for further scientific research and transparency, we must first evaluate internal policies, data protection regulations, and ethical considerations regarding participant privacy before determining a final plan.